CLINICAL TRIAL: NCT03951168
Title: Study on Standardized Management Model of Health Education for Diabetes Mellitus
Brief Title: Health Education for Diabetes Mellitus
Acronym: hefdm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018KRM115
Record Dates: First submitted 2019-05-04; First posted 2019-05-15 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Health education for diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Management (Other): The patients were divided into routine diabetic health education management model group. Patients who meet the criteria for admission and discharge.
  Interventions: Behavioral: Routine Management
- Standardized Management (Experimental): The patients were divided into standardized diabetes health education management model group. Patients who meet the criteria for admission and discharge.
  Interventions: Behavioral: Standardized Management

INTERVENTIONS:
Behavioral: Routine Management — Routine Management Model of Health Education for diabetes Patient will receive the Routine Management Model of Health Education for Diabetes. After the patient was admitted to hospital, the responsible nurse carried on the diabetes health education for the patient. There are no regulations on the path and time of education. Interspersed with diabetes health education at work. Follow up 2 weeks with phone call after discharge. This is the current clinical model in hospital.
  Arms: Routine Management
Behavioral: Standardized Management — Standardized Management Model of Health Education for Diabetes The patients were educated by full-time diabetic education nurses according to diabetes education path. Including diabetes diet, exercise, drugs, hypoglycemia, diabetic foot, and so on. Telephone follow-up was performed at 2 weeks and 4 weeks after discharge and 12 and 24 weeks follow-up in diabetes education clinic. Develop telephone follow-up standardized content and implement telephone follow-up according to standardized content.Full-time education nurses carry on education according to diabetes mellitus health education path table.
  Arms: Standardized Management

SUMMARY:
Through the construction and study of standardized diabetic health education management model. Routine diabetes health education management model was used in control group and standardized diabetes mellitus health education management model was used in intervention group. The changes of diabetic knowledge, self-management ability, quality of life,patient empowerment, HbA1c, and other metabolic indexes were observed.

DETAILED DESCRIPTION:
The aim was to develop a standardized patient education model reflecting the core educational elements recommended by Chinese diabetes society guideline, which could be delivered by nurses to hospitalized diabetes patients, and which could be easily scaled-up and implemented in China tier 3 hospital setting.

Management mode of standardized diabetes mellitus health education in intervention group.The control group carries on the routine diabetes mellitus health education management. In intervention group , All participants received Management mode of standardized diabetes mellitus health education.The standardized patient education included one-week personalized education on diabetes knowledge, diet and excise, glucose monitoring and hypoglycemia self-management and others during the hospitalization period. After discharge, patients were followed through the phone call at 2and 4 weeks. Follow-up of diabetic education outpatients at 12 and 24 weeks after discharge. The education nurse gave recommendations according to patent's problem during the follow-up. Full-time education nurses carry on education according to diabetes mellitus health education path table. In routine, After hospitalization, the responsible nurses interspersed with diabetes health education during the hospitalization. The health education is mainly about the problems observed by the responsible nurses and the problems raised by the patients. The patients were followed up by telephone 2 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients with World Health Organization(WHO) diagnosis (1999);
* HbA1c ≥ 7.5%;
* history of diabetes < 2 years;
* age from 18 to 70 years;
* having the ability of autonomous behavior, informed consent and voluntary participation in the study.

Exclusion Criteria:

* type 1 diabetes mellitus, gestational diabetes mellitus and other special types of diabetes;
* severe acute and chronic diseases, severe psychological failure, lung failure, tumor, etc.
* is participating in other researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Diabetes knowledge questionnaire ( DKQ) | after 6 months
  The DKQ was translated from English into Chinese by a native bilingual translation specialist and then back translated by a different native bilingual speaker and checked for accuracy, clarity and content equivalence by conducting forward and back translations to verify translation equivalence.
  DKQ was translated from English into Chinese by a native bilingual translation specialist and then back translated by a different native bilingual speaker and checked for accuracy,clarity and content equivalence by conducting forward and back translations to verify translation equivalence.
Summary of Diabetes Self-Care Activities-6 (SDSCA-6) | after 6 months
  Evaluation the patient self management skill
Diabetes empowerment Scale-Diabetes Attitudes Wishes & Needs Short Form (DES-DSF) | after 6 months
  Evaluation the patient empowerment
Diabetes Specific Quality of Life | after 6 months
  Evaluation the patient quality of life

SECONDARY OUTCOMES:
HbA1c | after 6 months
  the patient'S blood glucose level
Fasting glucose | after 6 months
  the patient'S blood glucose level
2h postprandial glucose | after 6 months
  the patient'S blood glucose level
blood pressure | after 6 months
  the patient 'S blood pressure
Total Cholesterol | after 6 months
  the patient'S Total Cholesterol
LDL-C | after 6 months
  he patient'S LDL-C
HDL-C | after 6 months
  he patient'S HDL-C

CONTACTS AND LOCATIONS:
Overall Officials: Meng Li, Study Chair — First Affiliated Hospital of Xi'an JiaoTong Univerisity
Locations (1):
- First affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No